CLINICAL TRIAL: NCT01965626
Title: A Multicenter Randomized Open-label Study of Oseltamivir Combined With High-dose Dexamethasone Versus High-dose Dexamethasone in the Management of Immune Thrombocytopenia
Brief Title: A Multicenter Randomized Open-label Study of Oseltamivir Combined With HD-DEX Versus HD-DEX in the Management of ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Oseltamivir; ITP-Oseltamivirphosphate (Registry Identifier: ITP-Oseltamivirphosphate)
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Thrombocytopenia
Keywords: Oseltamivir; Dexamethasone; ITP
MeSH Terms: conditions — Thrombocytopenia | interventions — Oseltamivir; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oseltamivir Combining HD-DXM (Active Comparator): Oseltamivir 75 mg twice per day, 10consecutive days
  HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Oseltamivir; Drug: Dexamethasone
- HD-DXM (Active Comparator): HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir 75 mg twice per day, 10 consecutive days
  Arms: Oseltamivir Combining HD-DXM
Drug: Dexamethasone — HD-DXM (orally at 40 mg daily for 4d)

SUMMARY:
Oseltamivirphosphate is hydrolysed to its active metabolite-the free carboxylate of oseltamivir. Oseltamivir is a neuraminidase inhibitor, serving as a competitive inhibitor of the activity of the viral neuraminidase (NA) enzyme upon sialic acid, found on glycoproteins on the surface of platelets. By blocking the activity of the enzyme, oseltamivir may prevent platelet destruction in liver.The project was undertaking by Qilu Hospital of Shandong University and other 4 well-known hospitals in China. In order to report the efficacy and safety of oseltamivirphosphate combined with high-dose dexamethasone for the treatment of immune thrombocytopenia (ITP) with high platelet desialylation level, compared to high-dose dexamethasone therapy.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 50 newly diagnosed ITP adult patients with high platelet desialylation level from 5 medical centers in China. One part of the participants are randomly selected to receiver HD-DXM (orally at 40 mg daily for 4d) combined with oseltamivir (orally at 75 mg twice for 10d), the others are selected to receive HD-DXM (orally at 40 mg daily for 4d ) alone. If platelet counts remained <30×109/L or there were bleeding symptoms by day 10, another 4-day course of HD-DXM was given (days 10-14).For the combination arm, patients with an initial response relapsed during the follow-up period, oseltamivir retreatment could be given for another 10 days at the discretion of the physician's advice and patients' will.

Platelet count, bleeding , platelet desialylation level and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of oseltamivirphosphate combining with high-dose dexamethasone therapy compared to high-dose dexamethasone for the treatment of adults with newly diagnosed ITP .

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ITP patients need of treatment(s) to minimize the risk of clinically significant bleeding primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* pregnancy hypertension cardiovascular disease diabetes liver and kidney function impairment HCV, HIV, HBsAg seropositive status patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
initial response and sustained response (SR) | Initial responses were assessed by day 14. Response lasting for at least 6 consecutive months without additional ITP-specific intervention was regarded as SR.
  CR: platelet count ≥ 100 × 109/L and absence of bleeding; R: platelet count ≥ 30 × 109/L but < 100 × 109/L and a doubling from baseline and absence of bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Derived] Sun L, Wang J, Shao L, Yuan C, Zhao H, Li D, Wang Z, Han P, Yu Y, Xu M, Zhao H, Qiu J, Zhou H, Liu X, Hou Y, Peng J, Hou M. Dexamethasone plus oseltamivir versus dexamethasone in treatment-naive primary immune thrombocytopenia: a multicentre, randomised, open-label, phase 2 trial. Lancet Haematol. 2021 Apr;8(4):e289-e298. doi: 10.1016/S2352-3026(21)00030-2. PMID 33770484